CLINICAL TRIAL: NCT01965912
Title: A Phase 4 Open-Label, Single-Cohort Study of the Long-Term Neurocognitive Outcomes in 4 to 5 Year-Old Children With Phenylketonuria Treated With Sapropterin Dihydrochloride (Kuvan®) for 7 Years
Brief Title: Kuvan®'s Effect on the Cognition of Children With Phenylketonuria
Acronym: KOGNITO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700773-002; 2009-015844-41 (EudraCT Number)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; Kuvan; Sapropterin dihydrochloride
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

ARMS (1):
- Kuvan® (Experimental)
  Interventions: Drug: Kuvan®

INTERVENTIONS:
Drug: Kuvan® — Kuvan® oral soluble tablet will be administered once daily along with Phenylalanine-restricted diet for a period of 7 years. Dosage of Kuvan® could range from 5 to 20 milligram per kilogram per day (mg/kg/day), as per Summary of Product Characteristics (SPC).
  Other Names: Sapropterin dihydrochloride

SUMMARY:
The study is a single-cohort, interventional, open-label trial to evaluate long-term neurocognitive (NC) outcomes in children aged 4 to 5 years with phenylketonuria (PKU) treated with Kuvan® and Phenylalanine-restricted diet over a period of 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients, 4 to 5 years of age (greater than or equal to 4 and less than 6) at the time of informed consent form signature by parent(s) or guardian(s)
* Confirmed clinical and biochemical diagnosis of PKU, including at least two separate blood phenylalanine levels greater than or equal to 400 micromole per liter (mcmol/L)
* Defined pre-Kuvan®/-tetrahydrobiopterin (BH4) dietary phenylalanine tolerance consistent with the diagnosis of PKU
* Responsive to Kuvan®/BH4:

  * For subjects currently treated with Kuvan®/BH4 at Screening: subject is a responder as per Investigator judgment based on documented effect of Kuvan®/BH4 on phenylalanine levels and/or phenylalanine tolerance
  * For subjects not treated with Kuvan®/BH4 at Screening: a response test has been performed during Screening or is available from the subject's medical records and satisfies the 3 following criteria: a decrease in blood phenylalanine levels of at least 30 percent was observed after at least 24 hours with a dose of at least 10 mg/kg/day
* Intelligence Quotient (IQ) greater than or equal to 70, as assessed with the Wechsler Preschool and Primary Scale of Intelligence (WPPSI)-III, 2nd part
* Good adherence with dietary treatment (including prescribed dietary phenylalanine restriction and prescribed amounts of phenylalanine-free protein supplements and low-phenylalanine foods), as assessed by the Investigator
* Well-controlled phenylalanine levels, as assessed by a minimum of 75 percent of phenylalanine levels within the target recommended in each centre during the previous 3 months
* Low phenylalanine diet started within the first 3 weeks of life
* Parent(s) or guardian(s) willing to comply with all study procedures, maintain strict adherence with the diet, and willing and able to provide written, signed informed consent before any trial-related activities are carried out, as well as ability of child to comply with trial procedures

Exclusion Criteria:

* Known hypersensitivity to Kuvan® or its excipients
* Known hypersensitivity to other approved or non-approved formulations of BH4
* Previous diagnosis of BH4 deficiency
* Current use of methotrexate, trimethoprim or other dihydrofolate reductase inhibitors
* Current use of medications that are known to affect nitric oxide synthesis, metabolism or action
* Current use of experimental or unregistered drugs (other than sapropterin/BH4) that may affect the study outcomes or use of such agents within 30 days prior to Screening
* Concurrent use of levodopa
* Concurrent disease or condition that would induce repeatedly catabolic situations, or interfere with the trial participation, diet, or NC development, as assessed by the Investigator
* Any condition that, in the view of the Investigator, renders the subject at high risk for failure to comply with treatment or to complete the trial
* Participation in a clinical trial investigating any other agent than Kuvan® within the past 30 days

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-10; Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Mean Full Scale Intelligence Quotient (FSIQ) Score of the Wechsler Intelligence Scale for Children (WISC)-IV | Year 7

SECONDARY OUTCOMES:
Height compared to the World Health Organization (WHO) Growth Standards | up to 7 years
Weight compared to the World Health Organization (WHO) Growth Standards | up to 7 years
Blood levels of tyrosine, tryptophan, pre-albumin and methylmalonic acid | up to 7 years
Intelligence Quotient (IQ) score and sub-scores such as, verbal IQ, performance IQ, Full Scale Intelligence Quotient (FSIQ) of Wechsler Preschool and Primary Scale of Intelligence (WPPSI)-III | Baseline
Intelligence Quotient (IQ) score and sub-scores such as verbal comprehension, perceptual reasoning, working memory, and processing speed indexes and Full Scale Intelligence Quotient (FSIQ) of the Wechsler Intelligence Scale for Children (WISC)-IV | up to 7 years
Change from Baseline in FSIQ score at 2, 4 and 7 years | Baseline, and Year 2, 4 and 7
Dietary Phenylalanine tolerance | up to 7 years
Phenylalanine levels | up to 7 years
Index of Dietary Control (IDC) | up to 7 years
Percentage of tablets taken to assess treatment compliance | up to 7 years
Distribution of phenylalanine hydroxylase (PAH) genotype | Baseline
Number of subjects with Adverse Events and Serious Adverse Events | up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Ece Kucuksayrac, MD, Study Director — BioMarin Pharmaceutical
Locations (12):
- Germany (2):
  - Research site, Munich
  - Research site, Münster
- Italy (3):
  - Research site, Bologna
  - Research site - Bambino Gesu, Roma
  - Research site - La Sapienza, Roma
- Spain (3):
  - Research Site, Barcelona
  - Research site, Murcia
  - Research site, Santiago de Compostela
- United Kingdom (4):
  - Research site, Birmingham
  - Research site, Bristol
  - Research Site - Evelina, London
  - Research site - GOSH, London